CLINICAL TRIAL: NCT04762056
Title: Validation of Chelsea Physical Assessment Tool (CPAx) in COVID-19 Patients for Assessing Functional Status After Intensive Care Unit Discharge
Brief Title: CPAx for Assessing Functional Status of COVID-19 Patients After Intensive Care Unit Discharge
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Post Intensive Care Unit Syndrome; Covid19
Keywords: post-intensive care syndrome; COVID-19; functional status; coronavirus
MeSH Terms: conditions — COVID-19; postintensive care syndrome; Coronavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients after ICU discharge: Patients who suffered COVID-19 pneumonia and stayed in ICU and discharged
  Interventions: Other: Chelsea Critical Care Physical Assessment Tool

INTERVENTIONS:
Other: Chelsea Critical Care Physical Assessment Tool — Chelsea Critical Care Physical Assessment Tool is a bedside assessment tool firstly reported in 2013 to measure physical morbidity in the critical care population, consisting of 10 items (respiratory function, cough, moving within the bed, supine to sitting on the edge of bed, dynamic sitting, standing balance, sit to stand, transferring from bed to chair, stepping, and grip strength) rated on a 6-point scale from complete dependency (level=0) to independency (level=5). Therefore, the CPAx sum score ranges from 0 (worst condition) to 50 (best functioning/independence)

SUMMARY:
The present assessment tools for assessing physical function after intensive care unit (ICU) can be categorized as (1) functional tests (2) walk tests (3) strength test (4) Health-related quality of life (HRQOL). Strength tests such as Medical Research Council Scale and HRQOL (e.g. Short form-36 (SF-36) tests may require awakening and appropriate mental health. However, mental impairments were seen in a considerable number of patients (2). Walk tests such as Six-Minute Walk Test (6MWT) or Timed Up&Go (TUG) can be impractical, some patients could not be able to perform these due to severe impairment. These tests require space to perform and may require management of several drips, drains, and oxygen delivery systems while the patient is walking and turning which render the test difficult to carry out. Among these three specific tools, CPAx seems to be the assessment tool that can be considered easy to use in the clinical setting due to the short time required for assessment and relatively minimal use of equipment (hand dynamometer for grip strength measurement).

This study aims to investigate validation of Chelsea Critical Care Physical Assessment Tool in the assessment of the functional status of COVID patients discharged from ICU and investigate the feasibility of commonly used assessment tools for assessing physical function after ICU in COVID patients discharged from ICU.

DETAILED DESCRIPTION:
The present assessment tools for assessing physical function after intensive care unit (ICU) can be categorized as (1) functional tests (2) walk tests (3) strength test (4) Health-related quality of life (HRQOL). Strength tests such as Medical Research Council Scale and HRQOL (e.g. SF-36) tests may require awakening and appropriate mental health. However, mental impairments were seen in a considerable number of patients (2). Walk tests such as Six-Minute Walk Test (6MWT) or Timed Up&Go (TUG) can be impractical, some patients could not be able to perform these due to severe impairment. These tests require space to perform and may require management of several drips, drains, and oxygen delivery systems while the patient is walking and turning which render the test difficult to carry out. Among functional tests, the Physical Function in Intensive Care Test (PFIT) Functional Status Score for the ICU and the Chelsea Critical Care Physical Assessment Tool (CPAx) are specifically designed to assess function after ICU while Barthel and Katz are nonspecific to this population. According to a systematic review of 26 different outcome measures, the CPAx and the Physical Function in Intensive Care Test demonstrated the strongest psychometric properties, however, the Physical Function in Intensive Care Test has a significant floor effect. The PFIT and CPAx may be more suitable for the assessment of patients who may never reach the ability to perform submaximal exercise tests.

Among these three specific tools, CPAx seems to be the assessment tool that can be considered easy to use in the clinical setting due to the short time required for assessment and relatively minimal use of equipment (hand dynamometer for grip strength measurement).

Patients over 18 years of age who suffered COVID-19 pneumonia and stayed in ICU and discharged will be included in the study. Patients who are able to follow at least 2 of the commands from De Jonghe and colleagues' awakening criteria will be evaluated within 48 hours discharge. Patients will be assessed by using Chelsea Critical Care Physical Assessment Tool, Barthel Index, Katz Index, 5 times Sit-To-Stand test, 30 seconds Sit-To-Stand test, Glasgow coma scale, handheld dynamometers, Medical Research Council sum score (MRC-SS) and modified Medical Research Council dyspnea scale. The number (%) of the patients who will be able to complete the tests will be recorded. Another physiatrist will also complete Chelsea Critical Care Physical Assessment Tool at the same time without discussion and will be blinded to score of the other rater. Patients' demographic characteristics such as age, gender, comorbidities will be recorded. Length of stay in ICU, duration of mechanical ventilation, history of Extra Corporeal Membrane Oxygenation (ECMO), presence of tracheostomy, intubation status, the sequential organ failure assessment score (SOFA score) at the day of ICU admission and acute physiology and chronic health evaluation (APACHE II) on ICU admission will be recorded.

For construct validation, the correlation between CPAx and Barthel, Katz, Medical Research Council sum score and grip strength will be calculated. Kappa and weighed Kappa analysis will be conducted for inter-rater reliability. Descriptive analysis (Number (%) of the patients who will be able to complete the tests) will be performed to assess feasibility.

This study aims to investigate validation of the Chelsea Critical Care Physical Assessment Tool in the assessment of the functional status of COVID patients discharged from ICU and investigate the feasibility of commonly used assessment tools for assessing physical function after ICU in COVID patients discharged from ICU.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (patients over 18 years of age)
2. Patients who suffered COVID-19 pneumonia and stayed in ICU and discharged. The patient will be assessed within 48 hours discharge
3. Patients who are able to follow at least 2 of the commands from De Jonghe and colleagues''(8) awakening criteria as follows:

Can patient follow the command? "Open/close your eyes." "Look at me." "Open your mouth and stick out your tongue." "Nod your head." "Raise your eyebrows when I have counted to 5."

Exclusion Criteria:

1. Patients with previous neurologic impairment
2. Pregnancy
3. Patients whose grip muscle strength cannot be evaluated (dominant extremity amputation etc.)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (patients over 18 years of age) who suffered COVID-19 pneumonia and stayed in ICU and discharged and who who are able to follow at least 2 of the commands from De Jonghe and colleagues' awakening criteria (presented below)
  De Jonghe and colleagues' awakening criteria
  Can patient follow the command? "Open/close your eyes." "Look at me." "Open your mouth and stick out your tongue." "Nod your head." "Raise your eyebrows when I have counted to 5."
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Chelsea Critical Care Physical Assessment Tool (CPAx) | Within 48 hours discharge
  The CPAx is a bedside assessment tool firstly reported in 2013 to measure physical morbidity in critical care population (12), consisting of 10 items (respiratory function, cough, moving within the bed, supine to sitting on the edge of bed, dynamic sitting, standing balance, sit to stand, transferring from bed to chair, stepping, and grip strength) rated on a 6-point scale from complete dependency (level=0) to independency (level=5), as depicted by Figure 1. Therefore, the CPAx sum score ranges from 0 (worst condition) to 50 (best functioning/independence)

SECONDARY OUTCOMES:
Barthel Index | Within 48 hours discharge
  The Barthel Scale/Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently following hospital discharge.Time taken and physical assistance required to perform each item are used in determining the assigned value of each item. The Barthel Index measures the degree of assistance required by an individual on 10 items of mobility and self care ADL. Proposed guidelines for interpreting Barthel scores are that scores of 0-20 indicate "total" dependency, 21-61 indicate "severe" dependency, 62-90 indicate "moderate" dependency, 91-99 indicates "slight" dependency, and 100 indicate ''full'' independent.
Katz Index | Within 48 hours discharge
  The Katz Index of Independence in Activities of Daily Living, commonly referred to as the Katz ADL, is the most appropriate instrument to assess functional status as a measurement of the client's ability to perform activities of daily living independently. Clinicians typically use the tool to detect problems in performing activities of daily living and to plan care accordingly. The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. Clients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Medical Research Council sum score (MRC-SS) | Within 48 hours discharge
  Medical Research Council (MRC)-sumscore evaluates global muscle strength. Manual strength of six muscle groups (shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, and ankle dorsiflexion) is evaluated on both sides using MRC scale. Summation of scores gives MRC-sumscore, ranging from 0 to 60. This score reliably identifies significant weakness (< 48) and even better in severe weakness (< 36) [4] which is the main medical interest for treatment in ICU-acquired weakness (ICUAW)
30 seconds sit to stand | Within 48 hours discharge
  The 30 Second Sit to Stand Test is also known as 30 second chair stand test ( 30CST), is for testing leg strength and endurance in older adults. It is part of the Fullerton Functional Fitness Test Battery. This test was developed to overcome the floor effect of the five or ten repetition sit to stand test in older adults.
5 times sit to stand test | Within 48 hours discharge
  The five Times Sit to Stand Test (5x Sit-To-Stand Test) commonly abbreviated as 5XSST is used to assesses functional lower extremity strength, transitional movements, balance, and fall risk in older adults
modified Medical Research Council (mMRC) dyspnea scale | Within 48 hours discharge
  The mMRC Dyspnea Scale quantifies disability attributable to breathlessness, and is useful for characterizing baseline dyspnea in patients with respiratory diseases. Describes baseline dyspnea, but does not accurately quantify response to treatment of chronic obstructive pulmonary disease (COPD).
Modified Borg scale | Within 48 hours discharge
  Borg rating of perceived exertion (RPE) is an outcome measure scale used in knowing exercise intensity prescription. It is use in monitoring progress and mode of exercise in cardiac patients as well as in other patient population undergoing rehabilitation and endurance training.
  Borg RPE scale was developed by Gunnar Borg for rating exertion and breathlessness during physical activity; that is, how hard the activity is as shown by high heart and respiration rate, profuse perspiration and muscle exertion.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Yilmaz Yalcinkaya, Prof, Study Director — Gaziosmanpasa Training and Research Hospital Physical and Rehabilitation Department; Zeynep Turan, MD, Study Chair — Koc University School of Medicine Department of Phsical Medicine and Rehabilitation; Mahir Topaloglu, MD, Study Chair — Koc University School of Medicine Department of Phsical Medicine and Rehabilitation; Ozden Ozyemisci Taskiran, Prof, Principal Investigator — Koc University School of Medicine Department of Phsical Medicine and Rehabilitation
Locations (2):
- Turkey (Türkiye) (2):
  - Deniz, Gaziosmanpaşa, Istanbul
  - Koç Univercity Hospital, Istanbul, None Selected

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study will be available on request from the corresponding author (EG). The data will not be publicly available due to their containing information that could compromise the privacy of research participants.

REFERENCES:
- [Result] Elliott D, Denehy L, Berney S, Alison JA. Assessing physical function and activity for survivors of a critical illness: a review of instruments. Aust Crit Care. 2011 Aug;24(3):155-66. doi: 10.1016/j.aucc.2011.05.002. Epub 2011 Jul 1. PMID 21723143
- [Result] Negrini F, Ferrario I, Mazziotti D, Berchicci M, Bonazzi M, de Sire A, Negrini S, Zapparoli L. Neuropsychological Features of Severe Hospitalized Coronavirus Disease 2019 Patients at Clinical Stability and Clues for Postacute Rehabilitation. Arch Phys Med Rehabil. 2021 Jan;102(1):155-158. doi: 10.1016/j.apmr.2020.09.376. Epub 2020 Sep 28. PMID 32991870
- [Result] Denehy L, de Morton NA, Skinner EH, Edbrooke L, Haines K, Warrillow S, Berney S. A physical function test for use in the intensive care unit: validity, responsiveness, and predictive utility of the physical function ICU test (scored). Phys Ther. 2013 Dec;93(12):1636-45. doi: 10.2522/ptj.20120310. Epub 2013 Jul 25. PMID 23886842
- [Result] Curci C, Pisano F, Bonacci E, Camozzi DM, Ceravolo C, Bergonzi R, De Franceschi S, Moro P, Guarnieri R, Ferrillo M, Negrini F, de Sire A. Early rehabilitation in post-acute COVID-19 patients: data from an Italian COVID-19 Rehabilitation Unit and proposal of a treatment protocol. Eur J Phys Rehabil Med. 2020 Oct;56(5):633-641. doi: 10.23736/S1973-9087.20.06339-X. Epub 2020 Jul 15. PMID 32667150
- [Result] Parry SM, Granger CL, Berney S, Jones J, Beach L, El-Ansary D, Koopman R, Denehy L. Assessment of impairment and activity limitations in the critically ill: a systematic review of measurement instruments and their clinimetric properties. Intensive Care Med. 2015 May;41(5):744-62. doi: 10.1007/s00134-015-3672-x. Epub 2015 Feb 5. PMID 25652888
- [Result] Holdar U, Eriksson F, Siesage K, Corner EJ, Ledstrom V, Svensson-Raskh A, Kierkegaard M. Cross-cultural adaptation and inter-rater reliability of the Swedish version of the Chelsea critical care assessment tool (CPAX-Swe) in critically ill patients. Disabil Rehabil. 2021 Jun;43(11):1600-1604. doi: 10.1080/09638288.2019.1668971. Epub 2019 Sep 26. PMID 31558043
- [Result] Nordon-Craft A, Schenkman M, Edbrooke L, Malone DJ, Moss M, Denehy L. The physical function intensive care test: implementation in survivors of critical illness. Phys Ther. 2014 Oct;94(10):1499-507. doi: 10.2522/ptj.20130451. Epub 2014 May 8. PMID 24810863
- [Result] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328